CLINICAL TRIAL: NCT01341340
Title: A Clinical Evaluation of the Everolimus Eluting Bioresorbable Vascular Scaffold System (BVS) for the Treatment of Subjects With Critical Limb Ischemia (CLI) From Occlusive Vascular Disease of the Tibial Arteries
Brief Title: The ABSORB BTK (Below The Knee) Clinical Investigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinued due to poor enrollment. Insufficient number of patients enrolled to permit a statistically rigorous assessment of safety and efficacy.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-112
Record Dates: First submitted 2011-04-15; First posted 2011-04-25 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Atherosclerosis; Peripheral Artery Disease; Peripheral Vascular Disease; PAD; Claudication; Critical Limb Ischemia; Lower Limb Disease; Peripheral Arterial Occlusive Disease; PAOD; PVD
Keywords: Stent; Infrapopliteal; Tibial; Limb Salvage
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease; Peripheral Vascular Diseases; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus Eluting BVS (Experimental): Patients receiving the Everolimus Eluting Bioresorbable Vascular Scaffold System (BVS)
  Interventions: Device: Everolimus Eluting BVS

INTERVENTIONS:
Device: Everolimus Eluting BVS — Patients receiving the Everolimus Eluting Bioresorbable Vascular Scaffold System (BVS)

SUMMARY:
The purpose of the ABSORB BTK Clinical Investigation is to evaluate the safety and efficacy of the Everolimus Eluting Bioresorbable Vascular Scaffold System (BVS) in subjects with critical limb ischemia (CLI) following percutaneous transluminal angioplasty (PTA) of the tibial arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 and ≤ 80 years of age.
2. History of symptomatic critical limb ischemia (CLI) (Rutherford Becker Clinical Category 4 or 5).
3. Subject is able to take at least one type of thienopyridine (e.g. clopidogrel) and acetylsalicylic acid (eg. Aspirin/ASA).
4. The subject must have a life-expectancy of more than 1 year.
5. Female subjects of childbearing potential must have had a negative pregnancy test within 14 days before treatment, must not be nursing at the time of treatment, and must also agree at time of consent to use birth control during participation in this study up to and including the angiographic follow-up at 1 year.
6. Subject has been informed of the nature of the study, agrees to its provisions, and has signed the informed consent form prior to any study related procedure.
7. Subject must agree to undergo all protocol-required follow-up examinations and requirements at the investigational site.
8. Subject must agree not to participate in any other clinical investigation for a period of one year following the index procedure. This includes clinical trials of medications and invasive procedures. Questionnaire-based studies, or other studies that are non-invasive and do not require medication are allowed.

Anatomic Inclusion Criteria

1. Up to two de novo lesions, each located in a separate native infrapopliteal vessel, with angiographically visible above-the-ankle reconstitution (proximal to the inferior cortical margin of the talus bone), only one of which can be designated as the target lesion and is suitable to be treated with a single BVS.
2. Target lesion length is visually estimated to be ≤ 24 mm.
3. Target vessel diameter at the location of the target lesion is ≥ 2.5 mm and ≤ 3.3 mm, as assessed by on-line quantitative angiography as per core laboratory guidelines.
4. The non-target lesion (if applicable) must be located in a separate infrapopliteal vessel, estimated to be ≤ 24 mm, and suitable to be treated with non-study percutaneous transluminal angioplasty (PTA) balloon(s) and/or a non-study stent.
5. Inflow between the proximal iliac and distal popliteal is unobstructed (free from ≥ 50% stenosis) as confirmed by angiography. [Note: Assessment may be made after interventions proximal to the target lesion.]
6. Subjects with a significant lesion (≥ 50% stenosis) in the inflow artery(ies) must have the inflow artery(ies) treated successfully prior to enrollment and treatment of the target lesion.
7. If there is evidence of an ischemic lesion/ulcer on the foot, the distribution of the target vessel must supply the area of the lesion (angiosome), as confirmed by angiography.
8. At least one patent distal tibial outflow artery (< 50% stenosis) that will provide a straight line of blood flow to the distal foot and (if applicable) wound area after treating a target lesion in the tibio-peroneal trunk.
9. Patent pedal outflow artery (< 50% stenosis) that will provide a straight line of blood flow to the distal foot and (if applicable) wound area.

Exclusion Criteria:

1. Subject is unable to understand or unwilling to cooperate with study procedures.
2. The subject is mentally ill or belongs to a vulnerable population.
3. Subject is currently breast-feeding, pregnant, or intends to become pregnant prior to completion of the 1 year angiographic follow-up.
4. Subject has had any type of amputation to the ipsilateral or contralateral extremity.
5. Subject is unable to walk. (with assistance is accepted)
6. Subject has had recent major surgery (requiring general or regional anesthesia or impacting major organ systems) within the last 3 months.
7. Subject has received, or is on the waiting list for a major organ transplant.
8. Subject is diagnosed as Rutherford Becker Clinical Category 0, 1, 2, 3 or 6.
9. Subject has any type of infection, until treated successfully.
10. Subject has osteomyelitis present in the distal ipsilateral extremity.
11. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
12. The subject has a history of prior life-threatening contrast media reaction.
13. Subject is receiving or scheduled to receive anticancer therapy for malignancy within 1 year prior to or after the procedure.
14. Subject is receiving immunosuppression therapy, or has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.).
15. Subject is receiving or will receive inhibitors of CYP3A or inducers of CYP3A within 30 days prior to or following the procedure.
16. Subject is receiving Phenprocoumon (Marcumar) or is scheduled to receive chronic anticoagulation therapy.
17. Subject has severe liver impairment as defined by total bilirubin > 3 mg/dl or two times increase over the normal level of serum glutamic oxaloacetic transminase(SGOT) or serum glutamic pyruvic transminase (SGPT).
18. Subject has platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC < 3,000 cells/mm3, or hemoglobin < 10.0 g/dl.
19. Subject has elevated serum creatinine > 2.0 mg/dl or > 150μmol/L.
20. Subject has uncontrolled diabetes mellitus (DM) (glucose > 400 mg/dl).
21. Subject has had a myocardial infarction (MI) within the previous 30 days or has unstable angina (defined as rest angina with ECG changes).
22. Subject has had a stroke within the previous 30 days and/or has deficits from a prior stroke that limits the subject's mobility.
23. Subject has acute thrombophlebitis or deep vein thrombosis in either extremity
24. Subject has known allergies to the following: aspirin, thienopyridines, heparin, contrast agent (that cannot be adequately treated with pre-medication or substitution for an alternate thienopyridine), poly (L-lactide), poly (DL-lactide), or drugs similar to everolimus (i.e. tacrolimus, sirolimus, zotarolimus), or other macrolides.
25. Subject requires any planned procedure that would necessitate the discontinuation of thienopyridines following the procedure. If the subject is enrolled into the study and then requires a medical procedure, which would necessitate the discontinuation of these medications, then the subject is to resume protocol recommended medications as soon as possible.
26. Subject has other known medical illnesses (e.g., cancer or congestive heart failure) that may cause the subject to be non-compliant with protocol requirements, confound the data interpretation, or is associated with limited life-expectancy (i.e., less than 1 year).
27. Subject is already participating in another clinical investigation that has not yet reached its primary endpoint.

Anatomic Exclusion Criteria

1. The target lesion can only be accessed via popliteal or pedal approach.
2. The target vessel diameter at the location of the target lesion is not suitable for available BVS size.
3. Unsuccessfully treated proximal inflow limiting arterial stenosis or inflow-limiting arterial lesions left untreated.
4. No angiographic evidence of a patent pedal artery.
5. Significant (> 50% stenosis) lesion in a distal outflow artery that requires treatment at the time of the index procedure.
6. More than a single significant lesion (> 50% stenosis) in the target vessel.
7. Target or (if applicable) non-target lesion location requiring bifurcation treatment method.
8. Target or (if applicable) non-target lesion lies within or adjacent to an aneurysm.
9. A segment/portion of the study scaffold will be deployed distal to the inferior cortical margin of the talus bone or in a pedal vessel.
10. Subject has previously had, or requires, bypass surgery, endarterectomy or other vascular surgery on any vessel of the ipsilateral extremity.
11. Subject has moderate to severe calcium in the target lesion or in the artery immediately adjacent to the target lesion, or the investigator is unable to pre-dilate the lesion according to vessel diameter.
12. Target or (if applicable) non-target vessel contains visible thrombus as indicated in the angiographic images.
13. Subject has angiographic evidence of thromboembolism or atheroembolism in the ipsilateral extremity. (Pre and post-angiographic images must confirm the absence of emboli in the distal anatomy.)
14. Target or (if applicable) non-target lesion has a high probability that a procedure other than pre-dilatation, implantation of the scaffold, and post-dilatation (as applicable) will be required at the time of index procedure for treatment of the target vessel (e.g., atherectomy, cutting balloon, etc.).
15. Subject has lesions in the target vessel that were treated or will require treatment < 1 year pre-or post- study procedure.
16. Subject has lesions in any other vascular anatomy, other than those treated at the time of the study procedure, that were treated or will require treatment < 30 days pre-or post- study procedure.
17. Subject has had or will require treatment with a drug-eluting/coated stent or drugcoated balloon in any vessel < 90 days pre-or post-study procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Freedom from major adverse limb events (MALE) within 1 year or peri-procedural (30-day) death (POD) (MALE+POD). | 1 year
  Major adverse limb events are defined as major amputations or major reinterventions. Major reinterventions include new bypass graft, jump/interposition graft revision, or thrombectomy /thrombolysis related to the target lesion, but do not include percutaneous endovascular reinterventions.

SECONDARY OUTCOMES:
Device Success | From start of index procedure to end of index procedure
  On a per device basis, the achievement of successful delivery and deployment of the study device(s) at the intended target lesion and successful withdrawal of the delivery catheter.
Technical Success | From start of index procedure to end of index procedure
  Defined on a per lesion basis, as the achievement of successful delivery and deployment of the study device(s) at the intended target lesion, successful withdrawal of the delivery catheter, and attainment of a final residual stenosis of < 30%.
Clinical Success | Within 48 hours after the index procedure or at hospital discharge, whichever is sooner
  On a per subject basis, technical success without complications within 48 hours after the index procedure or at hospital discharge, whichever is sooner.
Death | From start of procedure until discharge from treating or referral hospital
  all cause
Death | 1 month
  all cause.
Death | 6 months
  all cause.
Death | 1 year
  all cause.
Death | 2 years
  all cause.
Death | 3 years
  all cause.
Amputations | From start of procedure until discharge from treating or referral hospital
  minor and major
Amputations | 1 month
  minor and major
Amputations | 6 months
  minor and major
Amputations | 1 year
  minor and major
Amputations | 2 years
  minor and major
Amputations | 3 years
  minor and major
Limb Salvage | From start of procedure until discharge from treating or referral hospital
  Freedom from ipsilateral major amputations
Limb Salvage | 1 month
  Freedom from ipsilateral major amputations
Limb Salvage | 6 months
  Freedom from ipsilateral major amputations
Limb Salvage | 1 year
  Freedom from ipsilateral major amputations
Limb Salvage | 2 years
  Freedom from ipsilateral major amputations
Limb Salvage | 3 years
  Freedom from ipsilateral major amputations
Arterial thrombosis of the BVS | From start of procedure until discharge from treating or referral hospital
Arterial thrombosis of the BVS | 1 month
Arterial thrombosis of the BVS | 6 months
Arterial thrombosis of the BVS | 1 year
Arterial thrombosis of the BVS | 2 years
Arterial thrombosis of the BVS | 3 years
Amputation-free survival (AFS) | From start of procedure until discharge from treating or referral hospital
Amputation-free survival (AFS) | 1 month
Amputation-free survival (AFS) | 6 months
Amputation-free survival (AFS) | 1 year
Amputation-free survival (AFS) | 2 years
Amputation-free survival (AFS) | 3 years
Ipsilateral embolic events | From start of procedure until discharge from treating or referral hospital
Ipsilateral embolic events | 1 month
Ipsilateral embolic events | 6 months
Ipsilateral embolic events | 1 year
Ipsilateral embolic events | 2 years
Ipsilateral embolic events | 3 years
Freedom from target lesion revascularization (TLR)(ischemia driven and non-ischemia driven) | From start of procedure until discharge from treating or referral hospital
Freedom from target lesion revascularization (TLR)(ischemia driven and non-ischemia driven) | 1 month
Freedom from target lesion revascularization (TLR)(ischemia driven and non-ischemia driven) | 6 months
Freedom from target lesion revascularization (TLR)(ischemia driven and non-ischemia driven) | 1 years
Freedom from target lesion revascularization (TLR)(ischemia driven and non-ischemia driven) | 2 years
Freedom from target lesion revascularization (TLR)(ischemia driven and non-ischemia driven) | 3 years
Ipsilateral extremity revascularization (IER) | From start of procedure until discharge from treating or referral hospital
Ipsilateral extremity revascularization (IER) | 1 month
Ipsilateral extremity revascularization (IER) | 6 months
Ipsilateral extremity revascularization (IER) | 1 year
Ipsilateral extremity revascularization (IER) | 2 years
Ipsilateral extremity revascularization (IER) | 3 years
Peak Systolic Velocity Ratio (PSVR) | From start of procedure until discharge from treating or referral hospital
Peak Systolic Velocity Ratio (PSVR) | 1 month
Peak Systolic Velocity Ratio (PSVR) | 6 months
Peak Systolic Velocity Ratio (PSVR) | 1 year
Peak Systolic Velocity Ratio (PSVR) | 2 years
Peak Systolic Velocity Ratio (PSVR) | 3 years
Primary patency rate | From start of procedure until discharge from treating or referral hospital
Primary patency rate | 1 month
Primary patency rate | 6 months
Primary patency rate | 1 year
Primary patency rate | 2 years
Primary patency rate | 3 years
Secondary patency rate | From start of procedure until discharge from treating or referral hospital
Secondary patency rate | 1 month
Secondary patency rate | 6 months
Secondary patency rate | 1 year
Secondary patency rate | 2 years
Secondary patency rate | 3 years
Rutherford Becker clinical category and change from baseline for the treated limb | From start of procedure until discharge from treating or referral hospital
Rutherford Becker clinical category and change from baseline for the treated limb | 1 month
Rutherford Becker clinical category and change from baseline for the treated limb | 6 months
Rutherford Becker clinical category and change from baseline for the treated limb | 1 year
Rutherford Becker clinical category and change from baseline for the treated limb | 2 years
Rutherford Becker clinical category and change from baseline for the treated limb | 3 years
Ankle brachial index (ABI) and change from baseline for the treated limb | From start of procedure until discharge from treating or referral hospital
Ankle brachial index (ABI) and change from baseline for the treated limb | 1 month
Ankle brachial index (ABI) and change from baseline for the treated limb | 6 months
Ankle brachial index (ABI) and change from baseline for the treated limb | 1 year
Ankle brachial index (ABI) and change from baseline for the treated limb | 2 years
Ankle brachial index (ABI) and change from baseline for the treated limb | 3 years
Wound healing as measured by aggregate ulcer size and its change from baseline | From start of procedure until discharge from treating or referral hospital
Wound healing as measured by aggregate ulcer size and its change from baseline | 1 month
Wound healing as measured by aggregate ulcer size and its change from baseline | 6 months
Wound healing as measured by aggregate ulcer size and its change from baseline | 1 year
Wound healing as measured by aggregate ulcer size and its change from baseline | 2 years
Wound healing as measured by aggregate ulcer size and its change from baseline | 3 years
Walking capacity and change from baseline | From start of procedure until discharge from treating or referral hospital
Walking capacity and change from baseline | 1 month
Walking capacity and change from baseline | 6 months
Walking capacity and change from baseline | 1 year
Walking capacity and change from baseline | 2 years
Walking capacity and change from baseline | 3 years
Quality of Life Measures and change from baseline | From start of procedure until discharge from treating or referral hospital
Quality of Life Measures and change from baseline | 1 month
Quality of Life Measures and change from baseline | 6 months
Quality of Life Measures and change from baseline | 1 year
Quality of Life Measures and change from baseline | 2 years
Quality of Life Measures and change from baseline | 3 years
Target lesion mean and maximum treated site percent diameter stenosis (%DS) | 1 year
Target lesion mean treated site late loss | 1 year
Target lesion treated site binary restenosis | 1 year
Treated site Peak Systolic Velocity (PSV) | From start of procedure until discharge from treating or referral hospital
Treated site Peak Systolic Velocity (PSV) | 1 month
Treated site Peak Systolic Velocity (PSV) | 6 months
Treated site Peak Systolic Velocity (PSV) | 1 year
Treated site Peak Systolic Velocity (PSV) | 2 years
Treated site Peak Systolic Velocity (PSV) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Herz-Zentrum Leipzig
Locations (1):
- Abbott Vascular International Bvba, Diegem, Belgium